CLINICAL TRIAL: NCT02163902
Title: A Multicenter, Double-blind, Nontreatment, Long-term Follow up Study of Subjects Who Completed ATX-101 (Deoxycholic Acid Injection) Clinical Trials ATX-101-11-22 or ATX-101-11-23 for the Reduction of Localized Subcutaneous Fat in the Submental Area
Brief Title: Long-term Follow-up Study on Safety and Maintenance of Efficacy of ATX-101
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ATX-101-13-35
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Submental Fat; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATX-101 (Experimental): Participants treated with ATX-101 in previous studies ATX-101-11-22 and ATX-101-11-23.
  Interventions: Drug: ATX-101
- Placebo (Placebo Comparator): Participants treated with placebo in previous studies ATX-101-11-22 and ATX-101-11-23.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATX-101 — Clinical evaluation, patient reported outcome questionnaires, photographs, caliper measurements, recording of adverse events
  Arms: ATX-101
Drug: Placebo — Clinical evaluation, patient reported outcome questionnaires, photographs, caliper measurements, recording of adverse events
  Arms: Placebo

SUMMARY:
The investigation of the long-term safety and maintenance of efficacy of ATX-101 in reduction of submental fat.

DETAILED DESCRIPTION:
No study medication is administered in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Any participant who completed follow-up visits at 12 and 24 weeks after the last dose in one of the two predecessor studies
2. Willingness to comply with the schedule and procedures of this study.
3. Signed informed consent form (ICF).

Exclusion Criteria:

1. Participants who have had any treatment or condition (e.g., pregnancy or metabolic disease, which may lead to unstable weight) that may affect assessment of safety or efficacy since enrollment in the predecessor study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Beddingfield, III, MD, PhD, Study Director — Sponsor GmbH
Locations (15):
- United States (13):
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, San Diego, California
  - AboutSkin Dermatology and DermSurgery, PC, Englewood, Colorado
  - Dermatology Research Institute, Coral Gables, Florida
  - Stephan Baker MD PA, Coral Gables, Florida
  - Baumann Cosmetic and Research Center, Miami, Florida
  - Kenneth R. Beer, MD, PA, West Palm Beach, Florida
  - Altman Dermatology Associates, Arlington Hts, Illinois
  - DeNova Research, Chicago, Illinois
  - DuPage Medical Group, Dermatology Institute, Naperville, Illinois
  - Callender Center for Clinical Research, Glendale, Maryland
  - Aesthetics, Skin Care, Dermatologic Surgery, Rockville, Maryland
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Research Across America, Plano, Texas
- Canada (2):
  - Shannon Humphrey, MD, Vancouver
  - Carruthers Dermatology Centre Inc., Vancouver

REFERENCES:
- [Derived] Humphrey S, Cohen JL, Bhatia AC, Green LJ, Green JB, Bowen B. Improvements in Submental Contour up to 3 Years After ATX-101: Efficacy and Safety Follow-Up of the Phase 3 REFINE Trials. Aesthet Surg J. 2021 Oct 15;41(11):NP1532-NP1539. doi: 10.1093/asj/sjab100. PMID 33617632

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this non-treatment, double-blind, placebo-controlled follow-up study was to evaluate the long-term efficacy and safety of subcutaneous (SC) injections of deoxycholic acid (ATX-101) in the submental area. No treatment was administered in this study.
Pre-assignment Details: Participants who previously received deoxycholic acid or placebo injections in studies ATX-101-11-22 and ATX-101-11-23 were enrolled in this non-treatment, double-blind, placebo-controlled follow-up study to further evaluate safety and efficacy.
Groups:
- ATX-101 (Deoxycholic Acid) Injection: This is a non-treatment follow-up study. Participants were previously treated with deoxycholic acid injection, 10 mg/mL in 1 of 2 predecessor studies ATX-101-11-22 and ATX-101-11-23.
- Placebo: This is a non-treatment follow-up study. Participants were previously treated with placebo in 1 of 2 predecessor studies ATX-101- 11-22 and ATX-101-11-23.
Period: Overall Study
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Started | 113 | 111
Completed | 102 | 98
Not Completed | 11 | 13
Not completed — Subject's Request | 3 | 4
Not completed — Lost to Follow-up | 6 | 7
Not completed — Administrative Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo | Total
Number analyzed (Participants) | 113 | 111 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (8.22) | 50.1 (9.00) | 50.6 (8.61)
Age, Customized [Count of Participants; unit: Participants]
  ≤ 30 years | 3 | 4 | 7
  > 30 to ≤ 50 years | 52 | 49 | 101
  > 50 years | 58 | 58 | 116
  < 50 years | 47 | 47 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 95 | 191
  Male | 17 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 25 | 58
  Not Hispanic or Latino | 80 | 86 | 166
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 7 | 19
  White | 96 | 101 | 197
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.283 (4.4934) | 28.836 (4.0099) | 29.062 (4.2570)
Fitzpatrick Score [Count of Participants; unit: Participants] — Fitzpatrick skin type is a numerical classification schema for different skin types and tanning abilities. TYPE 1:
  Pale white skin, blue/hazel eyes, blond/red hair, always burns, never tans. TYPE 2: Fair skin, blue eyes, burns easily, tans poorly. TYPE 3: Darker white skin, tans after initial burn. TYPE 4: Light brown skin, burns minimally, tans easily. TYPE 5: Brown skin, rarely burns, tans darkly easily. TYPE 6: Dark brown or black skin, never burns, always tans darkly.
  Participants
    I | 4 | 4 | 8
    II | 30 | 39 | 69
    III | 33 | 36 | 69
    IV | 35 | 20 | 55
    V | 9 | 9 | 18
    VI | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining CR-SMFRS 1-Grade Response During 3 Years of Follow up, i.e. % of Participants Who Were CR-SMFRS 1-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: The investigator evaluated the participant's chin and neck area using the Clinician-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
  Non-responders at LTFU baseline in each treatment group (including placebo) were not included in the analysis.
Time Frame: From 12 weeks after last treatment (in the predecessor study) to up to 36 months after last treatment
Population: Participants who had at least a 1-grade reduction from baseline on the CRSMFRS (ie, CR-1 responder) at 12-weeks after last treatment in the predecessor studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 95 | 46
percentage of participants
  Visit 1 (Year 1) Percentage: number analyzed (Participants) | 88 | 44
  Visit 1 (Year 1) Percentage | 86.4 [79.2 to 93.5] | 56.8 [42.2 to 71.5]
  Visit 2 (Year 2) Percentage: number analyzed (Participants) | 85 | 42
  Visit 2 (Year 2) Percentage | 90.6 [84.4 to 96.8] | 73.8 [60.5 to 87.1]
  Visit 3 (Year 3) Percentage: number analyzed (Participants) | 85 | 40
  Visit 3 (Year 3) Percentage | 82.4 [74.2 to 90.5] | 65.0 [50.2 to 79.8]

2. Secondary Outcome: Percentage of Participants Maintaining CR-SMFRS 2-Grade Response During 3 Years of Follow up, i.e. % of Participants Who Were CR-SMFRS 2-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: as for outcome 1
Time Frame: From 12 weeks after last treatment (in the predecessor study) to up to 36 months after last treatment.
Population: Analysis Population: Participants who had at least a 2-grade reduction from baseline on the CR-SMFRS (ie, CR-2 responder) at 12-weeks after last treatment in the predecessor studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 44 | 12
percentage of participants
  Visit 1 (Year 1) Percentage: number analyzed (Participants) | 40 | 11
  Visit 1 (Year 1) Percentage | 75.0 [61.6 to 88.4] | 18.2 [0.0 to 41.0]
  Visit 2 (Year 2) Percentage: number analyzed (Participants) | 40 | 9
  Visit 2 (Year 2) Percentage | 72.5 [58.7 to 86.3] | 33.3 [2.5 to 64.1]
  Visit 3 (Year 3) Percentage: number analyzed (Participants) | 38 | 9
  Visit 3 (Year 3) Percentage | 65.8 [50.7 to 80.9] | 33.3 [2.5 to 64.1]

3. Secondary Outcome: Percentage of Participants Maintaining PR-SMFRS 1-Grade Response During 3 Years of Follow up, i.e. % of Participants Who Were PR-SMFRS 1-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: The participant evaluated their chin and neck area using the Patient-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
  Non-responders at LTFU baseline in each treatment group (including placebo) were not included in the analysis.
Time Frame: From 12 weeks after last treatment (in the predecessor study) to up to 36 months after last treatment
Population: Analysis Population: Participants who had at least a 1-grade reduction from baseline in PR-SMFRS (ie, PR-1 responder) at 12-weeks after last treatment in the predecessor studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 98 | 58
percentage of participants
  Visit 1 (Year 1) Percentage: number analyzed (Participants) | 88 | 55
  Visit 1 (Year 1) Percentage | 95.5 [91.1 to 99.8] | 76.4 [65.1 to 87.6]
  Visit 2 (Year 2) Percentage: number analyzed (Participants) | 90 | 53
  Visit 2 (Year 2) Percentage | 87.8 [81.0 to 94.5] | 83.0 [72.9 to 93.1]
  Visit 3 (Year 3) Percentage: number analyzed (Participants) | 87 | 48
  Visit 3 (Year 3) Percentage | 77.0 [68.2 to 85.9] | 75.0 [62.8 to 87.2]

4. Secondary Outcome: Percentage of Participants Maintaining PR-SMFRS 2-Grade Response During 3 Years of Follow up, i.e. % of Participants Who Were PR-SMFRS 2-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: as for outcome 3
Time Frame: From 12 weeks after last treatment (in the predecessor study) to up to 36 months after last treatment
Population: Analysis Population: Participants who had at least a 2-grade reduction from baseline in PR-SMFRS (ie, PR-2 responder) at 12-weeks after last treatment in the predecessor studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 43 | 11
percentage of participants
  Visit 1 (Year 1) Percentage: number analyzed (Participants) | 39 | 11
  Visit 1 (Year 1) Percentage | 59.0 [43.5 to 74.4] | 63.6 [35.2 to 92.1]
  Visit 2 (Year 2) Percentage: number analyzed (Participants) | 40 | 10
  Visit 2 (Year 2) Percentage | 57.5 [42.2 to 72.8] | 60.0 [29.6 to 90.4]
  Visit 3 (Year 3) Percentage: number analyzed (Participants) | 37 | 10
  Visit 3 (Year 3) Percentage | 59.5 [43.6 to 75.3] | 70.0 [41.6 to 98.4]

5. Secondary Outcome: Percentage of Participants Maintaining Composite SMFRS 1-Grade Response During 3 Years of Follow up, i.e. % of Participants Who Were CR-SMFRS and PR-SMFRS 1-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: The investigator evaluated the participant's chin and neck area using the Clinician-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=absent submental convexity (best) to 4= extreme submental convexity (worst).
  The participant evaluated their chin and neck area using the Patient-Reported Submental Fat Rating Scale (a 5-point scale) where: 0=no chin fat at all (best) to 4= a very large amount of chin fat (worst).
  Non-responders at LTFU baseline in each treatment group (including placebo) were not included in the analysis.
Time Frame: From 12 weeks after last treatment (in the predecessor study) to up to 36 months after last treatment
Population: Analysis Population: Participants who were both CR-1 responders and PR-1 responders (SMFRS-1) at 12-weeks after last treatment in the predecessor studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 83 | 31
percentage of participants
  Visit 1 (Year 1) Percentage: number analyzed (Participants) | 76 | 29
  Visit 1 (Year 1) Percentage | 86.8 [79.2 to 94.4] | 44.8 [26.7 to 62.9]
  Visit 2 (Year 2) Percentage: number analyzed (Participants) | 74 | 28
  Visit 2 (Year 2) Percentage | 85.1 [77.0 to 93.2] | 64.3 [46.5 to 82.0]
  Visit 3 (Year 3) Percentage: number analyzed (Participants) | 73 | 26
  Visit 3 (Year 3) Percentage | 72.6 [62.4 to 82.8] | 46.2 [27.0 to 65.3]

6. Secondary Outcome: Percentage of Participants Maintaining Composite SMFRS 2-Grade Response During 3 Years of Follow up, i.e. % of Participants Who Were CR-SMFRS and PR-SMFRS 2-Grade Responders at Both Long-term LTFU Baseline and at Subsequent LTFU Visits
Description: as for outcome 5
Time Frame: From 12 weeks after last treatment (in the predecessor study) to up to 36 months after last treatment
Population: Analysis Population: Participants who were both CR-2 responders and PR-2 responders (SMFRS-2) at 12-weeks after last treatment in the predecessor studies.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
Number analyzed (Participants) | 18 | 3
percentage of participants
  Visit 1 (Year 1) Percentage: number analyzed (Participants) | 17 | 3
  Visit 1 (Year 1) Percentage | 41.2 [17.8 to 64.6] | 0.0 [NA to NA] — Of the 3 SMFRS-2 responders in the Placebo group 0 participants maintained response.
  Visit 2 (Year 2) Percentage: number analyzed (Participants) | 16 | 2
  Visit 2 (Year 2) Percentage | 43.8 [19.4 to 68.1] | 0.0 [NA to NA] — Of the 3 SMFRS-2 responders in the Placebo group 0 participants maintained response.
  Visit 3 (Year 3) Percentage: number analyzed (Participants) | 14 | 2
  Visit 3 (Year 3) Percentage | 50.0 [23.8 to 76.2] | 50.0 [0.0 to 100.0]

ADVERSE EVENTS:
Time Frame: From the first exposure to study drug in predecessor study to up to 36 months after last treatment in predecessor study
Description: All enrolled participants with a clearly identifiable actual treatment received from a previous ATX-101 study and at least 1 visit in the long-term follow-up (LTFU) study were included in the analysis population. All adverse events (AEs) and serious adverse events (SAEs) that were ongoing at the conclusion of the predecessor Studies ATX-101-11-22 and ATX-101-11-23 were followed until they resolved or were considered medically stable.
Arm/Group | ATX-101 (Deoxycholic Acid) Injection | Placebo
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/111
Serious Adverse Events (participants affected / at risk) | 5/113 | 1/111
Other Adverse Events (participants affected / at risk) | 0/113 | 0/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ATX-101 (Deoxycholic Acid) Injection (N=113) | Placebo (N=111)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Breast reconstruction (Surgical and medical procedures) | 1/96 (1) | 0/95 (0)
Ovarian cancer recurrent (Reproductive system and breast disorders) | 1/96 (1) | 0/95 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/96 (0) | 1/95 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.